CLINICAL TRIAL: NCT05650983
Title: Effect of Exercise on Cognitive Function and Mental Health in Heroin Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Sport University (Other)
Responsible Party: Principal Investigator, Chunlu Fang, Principal Investigator, Guangzhou Sport University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022LcLL-30
Record Dates: First submitted 2022-11-08; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Unspecified Symptoms and Signs Involving Cognitive Functions Following Unspecified Cerebrovascular Disease; Heroin Addicts; Executive Function; Negative Thinking/Affect
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.Aerobic exercise (Experimental): play balloon volleyball for Aerobic exercise and aimed at maximizing the strain on the cardiovascular system (60-70% of heart rate recovery). Aerobic exercise intervention five times a week, one hour each time，for three months.
  Interventions: Behavioral: Aerobic exercise; Resistance exercise
- 2.Resistance exercise (Experimental): Resistance strength training for Resistance exercise and aimed at promoting the greatest hypertrophy response(65% of 1 repetition maximum and repeated up to 15 times). Resistance exercise intervention five times a week, one hour each time,for three months.
  Interventions: Behavioral: Aerobic exercise; Resistance exercise

INTERVENTIONS:
Behavioral: Aerobic exercise; Resistance exercise — To investigate affect/effect of dissimilar modes of exercise, Aerobic exercise versus Resistance exercise, on execution function and psychological symptoms in heroin addicts, 1 hour of characteristic exercise protocols aiming to (a) maximize the strain on the cardiovascular system with Aerobic exercise(60-70% of heart rate recovery) and (b) promote the greatest hypertrophy response with Resistance exercise(65% of 1 repetition maximum & repeated up to 15 time) were used. Both exercise programs were designed to match the male heroin addicts, with medium-intensity Strength-Trained for Resistance exercise and playing balloon volleyball for Aerobic exercise. Two exercise groups performed at 65% of their pre-determine peak oxygen uptake.

SUMMARY:
The goal of this [type of study: exercise intervention study] is to test in describe participant health conditions. The main questions it aims to answer are:

* [Whether physical exercise improves executive function of male heroin addicts]
* [Whether physical exercise improves negative thinking/affect psychological experience of male heroin addicts] Participants will be randomly selected for medium-intensity strength training (resistance exercise,n=30), 30 will be selected for 1-hour long balloon volleyball sessions (aerobic exercise) at 60-70% volume of oxygen uptake during peak exercise, weekly 5 times for 12 weeks; and 30 will be assigned to the no-exercise control group, Participants will perform Executive function tests and the Symptom Checklist-90 Revised questionnaire at pre and post intervention.

Researchers will compare resistance exercise group,aerobic exercise group and no-exercise control group to see if effects of exercise on executive function and negative thinking/affect psychological experience of male heroin addicts.

ELIGIBILITY:
Inclusion Criteria:

* were men who met the Manual of Mental Disorders (DSM)-IV criteria for current heroin dependence

Exclusion Criteria:

* any major mental illness other than heroin addiction
* any exercise taboo

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
using the Symptom Checklist-90-R (SCL-90-R) questionnaire to investigate the improvement of physical exercise on psychological symptoms in heroin addicts, | Month 3
  Participants will be assessed the Symptom Checklist-90-R (SCL-90-R) questionnaire at pre and post exercise intervention.
using the executive functioning tests to investigate the improvement of physical exercise on executive function in heroin addicts, | Month 3
  Participants will perform executive function test

CONTACTS AND LOCATIONS:
Locations (1):
- Desk and Computer and Playground, Guangzhou, Guangdongsheng, China

IPD SHARING:
Plan to Share IPD: No